CLINICAL TRIAL: NCT03048526
Title: Influence of Perfluorohexyloctane (NovaTears) on Tear Film Thickness in Patients With Mild to Moderate Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novaliq GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NT-004
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NovaTears® (Experimental)
  Interventions: Device: NovaTears®
- Hydrabak® (Active Comparator): Unpreserved sodium chloride (0.9%) eye drops in ABAK® system
  Interventions: Device: Hydrabak®

INTERVENTIONS:
Device: NovaTears® — Topical eye drops for lubrication of the ocular surface
  Arms: NovaTears®
Device: Hydrabak® — Eye drops
  Arms: Hydrabak®

SUMMARY:
Patients with mild to moderate dry eye disease will be randomized to receive either NovaTears® or Hydrabak® eye drops as control.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* History of dry eye disease for at least 3 months before the screening visit
* Be able and willing to follow instructions, including participation in all study assessments and visits
* Signed and dated written informed consent

Exclusion Criteria:

* Have any clinically significant slit-lamp findings at the screening visit that may include trauma, Steven Johnson syndrome, and/or in the opinion of the investigator may interfere with study parameters
* Participation in a clinical trial in the 4 weeks preceding the before the screening visit
* Active ocular allergies or ocular allergies that are expected to be active during the study period
* Pregnancy, planned pregnancy or lactating
* Known hypersensitivity to any component of the study medication
* Any medical or surgical history, disorder or disease such as acute or chronic severe organic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
Tear film thickness as measured with high resolution optical coherence tomography | 4 weeks

SECONDARY OUTCOMES:
Lipid layer thickness | 4 weeks
Non-invasive tear break up time | 4 weeks
Dynamic Meibomian Gland Imaging | 4 weeks
Blink frequency | 4 weeks
Symptom VAS | 4 weeks
Corneal fluorescein staining | 4 weeks
Conjunctival lissamine green staining | 4 weeks
Schirmer I test | 4 weeks
Tear film break up time | 4 weeks
Ocular surface disease index | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhoefer, MD, Study Director — Novaliq GmbH
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Austria